CLINICAL TRIAL: NCT01247324
Title: A Randomized, Double-Blind, Double-Dummy, Parallel-Group Study To Evaluate the Efficacy and Safety of Ocrelizumab in Comparison to Interferon Beta-1a (Rebif®) in Patients With Relapsing Multiple Sclerosis
Brief Title: A Study of Ocrelizumab in Comparison With Interferon Beta-1a (Rebif) in Participants With Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA21092; 2010-020337-99 (EudraCT Number)
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — Interferon beta-1a; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interferon beta-1a 44 mcg SC (Active Comparator): Interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).
  Interventions: Drug: Interferon beta-1a; Drug: Ocrelizumab-matching placebo
- Ocrelizumab (Experimental): Ocrelizumab 600 mg intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week.
  Interventions: Drug: Ocrelizumab; Drug: Interferon beta-1a-matching placebo

INTERVENTIONS:
Drug: Interferon beta-1a
  Other Names: Rebif
  Arms: Interferon beta-1a 44 mcg SC
Drug: Ocrelizumab-matching placebo
  Arms: Interferon beta-1a 44 mcg SC
Drug: Ocrelizumab
  Other Names: RO4964913
  Arms: Ocrelizumab
Drug: Interferon beta-1a-matching placebo
  Arms: Ocrelizumab

SUMMARY:
This randomized, double-blind, double-dummy, parallel-group study will evaluate the efficacy and safety of ocrelizumab in comparison with interferon beta-1a (Rebif) in participants with relapsing multiple sclerosis. Participants will be randomized to receive either ocrelizumab 600 mg or matching placebo intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week; or interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks). Planned duration of double-blind treatment is 96 weeks. Participants who complete the 96-week double-blind treatment will have an option to enter a single-group, active-treatment, open-label extension period, providing they fulfill the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis, in accordance with the revised McDonald criteria (2010)
* At least 2 documented clinical attacks within the last 2 years prior to screening or one clinical attack in the years prior to screening (but not within 30 days prior to screening)
* Neurologic stability for greater than or equal to (>=) 30 days prior to both screening and baseline
* Expanded Disability Status Scale (EDSS) score 0 to 5.5 inclusive

Exclusion Criteria:

* Primary progressive multiple sclerosis
* Disease duration of more than 10 years in participants with EDSS less than or equal to (<=) 2.0 at screening
* Contraindications for MRI
* Known presence of other neurological disorders which may mimic multiple sclerosis
* Pregnancy or lactation
* Requirement for chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* History of or currently active primary or secondary immunodeficiency
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Active infection, or history of or known presence of recurrent or chronic infection (e.g., hepatitis B or C, human immunodeficiency virus [HIV], syphilis, tuberculosis)
* History of progressive multifocal leukoencephalopathy
* Contraindications to or intolerance of oral or iv corticosteroids
* Contraindications to Rebif or incompatibility with Rebif use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 821 (Actual)
Dates: Start 2011-08-31 (Actual); Primary Completion 2015-04-02 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (142):
- United States (40):
  - 21st Century Neurology, Phoenix, Arizona
  - Mercy Medical Group, Carmichael, California
  - Scripps Clinic, La Jolla, California
  - MS Center of California, Laguna Hills, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Neuro-Therapeutics Inc., Pasadena, California
  - University of California at San Francisco, San Francisco, California
  - Health First Physicians Inc., Melbourne, Florida
  - Mercy Research Institute, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Shepherd Center Inc., Atlanta, Georgia
  - Emory University; Department of Neurology, Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Northwestern University; Dept. of Neurology, Chicago, Illinois
  - Consultants in Neurology Ltd, Northbrook, Illinois
  - American Health Network Institute, LLC, Avon, Indiana
  - Massachusetts General Hospital., Boston, Massachusetts
  - Michigan Neurology Associates P.C., Clinton Township, Michigan
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - The Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - The MS Center for Innovations In Care, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - The MS Center; Advance Neurology and Pain, Advance, North Carolina
  - Atrium Health Neurosciences Institute ? Charlotte, Charlotte, North Carolina
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Neurology Associates PA, Hickory, North Carolina
  - University Neurology Inc., Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Providence Neurological Specialties, Portland, Oregon
  - Albert Einstein Medical Center; Depatment of Neurosensory sciences, Philadelphia, Pennsylvania
  - Magee-Woman's Hospital, Pittsburgh, Pennsylvania
  - Uni of Texas Health Science Center At Houston, Houston, Texas
  - Bhupesh Dihenia M.D. P.A., Lubbock, Texas
  - Uni of Vermont Medical Center;, Burlington, Vermont
  - Multicare Research Institute; Multicare Neuroscience Center of Washington, Tacoma, Washington
- Argentina (3):
  - Instituto centenario, Buenos Aires
  - Hospital Español, Ciudad Autonoma Bs As
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
- Royal North Shore Hospital; Department of Neurology, St Leonards, New South Wales, Australia
- Barmherzige Brueder Konventspital, Linz, Austria
- Belgium (3):
  - AZ Sint Jan, Bruges
  - Cliniques Universitaires Saint-Luc; Neurology, Brussels
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (3):
  - Hospital das Clinicas - UFG;Reumatologia, Goiânia, Goiás
  - IMV Pesquisa Neurológica, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica; Neurocirurgica de Joinville, Joinville, Santa Catarina
- Bulgaria (5):
  - MHAT Avis Medica; Neurology Department, Pleven
  - First MHAT; Clinic of Neurology, Sofia
  - MHATNP Sv.Naum EAD; Clinic in neurology diseases for movement disorders, Sofia
  - ACIBADEM CITY CLINIC TOKUDA HOSPITAL EAD; Clinic of Neurology and Sleep Medicine, Sofia
  - Military Medical Academy; Neurology, Sofia
- Hospital Carlos Van Buren, Valparaíso, Chile
- Czechia (6):
  - Fakultni nemocnice u sv. Anny; Neurologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava; NEU-Neurologicke oddeleni, Jihlava
  - Krajska Nemocnice Pardubice Neurologicka Klinika, Pardubice
  - VFN Praha Poliklinika Rs Centrum - Budova A, Prague
  - Krajska zdravotni, a. s. ? Nemocnice Teplice, o. z.; Neurologicke oddeleni, Teplice
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- FinnMedi Oy, Tampere, Finland
- France (5):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Hopital Gabriel Montpied; Service de Neurologie, Clermont-Ferrand
  - Hopital Central; Neurologie, Nancy
  - CHU de Nîmes Hopital Caremeau; Service de Neurologie, Nîmes
  - Hopital Hautepierre - CHU Strasbourg; Service de Neurologie, Strasbourg
- Germany (10):
  - Charité Universitaetsmedizin Berlin, Campus Charité Mitte, Berlin
  - Universitätsklinikum "Carl Gustav Carus"; MS Center Dresden, Dresden
  - Asklepiosklinik Barmbek; Abteilung Neurologie, Hamburg
  - Diakoniekrankenhaus Henriettenstiftung gGMBH; Klinik für Neurologie und klinische Neurophysiologie, Hanover
  - Universitaetsklinikum Mainz - PS; Klinik und Poliklinik fuer Neurologie, Mainz
  - Praxis Dr. med. Mathias Niedhammer, Facharzt für Neurologie, Oldenburg
  - Neurozentrum Prien Elisabeth Hans-Thümmler Stefan Braune, Prien am Chiemsee
  - Universitätsklinikum Rostock, Zentrum für Nervenheilkunde; Klinik und Poliklinik für Neurologie, Rostock
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Studienzentrum Nordwest Dr med Joachim Springub Herr Wolfgang Schwarz, Westerstede
- Hungary (3):
  - Semmelweis Egyetem AOK; Neurologiai Klinika, Budapest
  - Fovarosi Onkormanyzat Jahn Ferenc Del-Pesti, Budapest
  - Szent Borbala Korhaz; Neurology, Tatabánya
- Chaim Sheba Medical Center; Neurology Department, Ramat Gan, Israel
- Italy (4):
  - Azienda Socio Sanitaria Territoriale della Valle Olona (pres, Gallarate, Aosta Valley
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Azienda Ospedaliera di Padova; Clinica Neurologica, Padua, Veneto
- Latvia (2):
  - Maritime Medicine Centre of Latvia Hospital of Vecmilgravis Department of Neurology, Riga
  - P. Stradins Clinical University Hospital; Neurology, Riga
- Lithuania (3):
  - Kaunas Medical University Hospital, Kaunas
  - Klaipeda University Hospital Public Institution, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Vilnius
- Mexico (2):
  - Grupo Médico Camino S.C., Mexico City, Mexico CITY (federal District)
  - Hospital Universitario Dr Jose Eleuterio Gonzalez; Universidad Autónoma de Nuevo León, Monterrey, Nuevo León
- St. Antonius Ziekenhuis Nieuwegein, Nieuwegein, Netherlands
- Peru (4):
  - Policlinico Especializado en Neurologia, Callao
  - Clinica Anglo Americana, Lima
  - Hospital Nacional Dos de Mayo, Lima
  - Clinica Centenario Peruano Japonesa; Neurology, Pueblo Libre
- Poland (4):
  - COPERNICUS Podmiot Leczniczy Sp. z o. o. Szpital im. M. Kopernika; Oddzia? Neurologiczny, Gdansk
  - Specjal. Praktyka Lekarska; Prof. Grzegorz Opala, Katowice
  - MA-LEK Clinical Sp. Z o.o., Katowice
  - Neurologiczny NZOZ Centrum Leczenia SM; Osrodek Badan Klinicznych, Plewiska
- Hospital de Braga; Servico de Neurologia, Braga, Portugal
- Russia (12):
  - Central Clinical Hospital #2 N.A. Semashko OAO RJHD, Moskva, Moscow Oblast
  - FGBU FNKC FMBA of Russia, Moskva, Moscow Oblast
  - MMA of Ministry of Defense of Russia named after S.M. Kirov, Saint Petersburg, Sankt-Peterburg
  - St.-Peterburg State institution of health care City multifield hospital #2, Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg, Sverdlovsk Oblast
  - Regional Multiple Sclerosis Centre b/o CC ECM "Neftyanik", Tyumen, Tyumen Oblast
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - FSBIH Siberian Regional Medical Centre of FMBA of Russia, Novosibirsk
  - MRC for Oncology and Neurology Biotherapy, Novosibirsk
  - Samara State Medical University, Samara
  - Reg. SI of Health Care Smolensk Regional Clinical Hospital, Smolensk
  - Regional Multiple Sclerosis Centre b/o CC ECM "Neftyanik", Tyumen
- Serbia (3):
  - Military Medical Academy, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- Slovakia (4):
  - FNsP Bratislava - Nemocnica Stare mesto, Bratislava
  - FNsP Bratislava, Nemocnica Ruzinov, Bratislava
  - Univerzitna nemocnica Bratislava Nemocnica sv. Cyrila a Metoda; Nemocnicna lekaren, Bratislava
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- Dr CC Coetzee Inc, Durban, South Africa
- Spain (4):
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Neurologia, Santa Cruz de Tenerife, Tenerife
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitario Puerta De Hierro Majadahonda; Servicio de Neurología, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- Switzerland (2):
  - Universitätsspital Basel Medizin Neurologie; Neurologische Poliklinik, Basel
  - Ospedale Regionale Lugano Civico Medizin Neurologie; Neurologia, Lugano
- Tunisia (3):
  - Hopital Razi, Mannouba
  - Hopital Universitaire Fattouma Bourguiba, Monastir
  - Hopital Charles Nicolle, Tunis
- Ukraine (5):
  - MMPIDon.Reg.Cl.&Ter.Med.Com.Neur.Dept.DNMU n.a.M.Gorkiy; Ch. of Nervous Diseases and Med. Genetics, Donetsk
  - St.In.Inst. of Neurol.Psych.and Narcol.of the AMSU; Dept. of Neuroinfection and Multiply Sclerosis, Kharkiv
  - Kyiv City Cl.Hosp.#4 Depart.of Neurology #2NMU; Department of Neurology, Kyiv
  - Lviv Regional Clinical Hospital; Department of Neurology, Lviv
  - Vin.Reg.Psych.Hosp.N.A Yuschenko O.I., Vnmu N.A. Pyrogov; Department of Nervous Diseases, Vinnytsia
- United Kingdom (2):
  - Walton Centre NHS Foundation Trust, Neuroscience Research Centre; CLINICAL TRIALS UNIT, Liverpool
  - Royal London Hospital; Neurology, London

REFERENCES:
- [Derived] Kappos L, Yiu S, Reucassel J, Oh J, Granziera C, Killestein J, Bermel RA, Berge C, Kazlauskaite A, Schneble HM, Dahlke F, Cree BAC. Performance of Composite Endpoints Defining Progression Independent of Relapse Activity in Multiple Sclerosis. Ann Clin Transl Neurol. 2025 Sep;12(9):1805-1812. doi: 10.1002/acn3.70111. Epub 2025 Jul 8. PMID 40629721
- [Derived] Montobbio N, Bovis F, Signori A, Carmisciano L, Schiavetti I, Ponzano M, Tur C, Granziera C, Cagol A, Arnold DL, Kappos L, Sormani MP. Uncovering a bias in estimated treatment effects on PIRA in multiple sclerosis clinical trials. EBioMedicine. 2025 Jul;117:105802. doi: 10.1016/j.ebiom.2025.105802. Epub 2025 Jun 18. PMID 40554392
- [Derived] Kappos L, Yiu S, Dahlke F, Coetzee T, Cutter GR, Yuen S, Bonati U, Lublin FD. Composite Confirmed Disability Worsening/Progression Is a Useful Clinical Endpoint for Multiple Sclerosis Clinical Trials. Neurology. 2025 May 27;104(10):e213558. doi: 10.1212/WNL.0000000000213558. Epub 2025 Apr 21. PMID 40258203
- [Derived] Benedict RH, Kappos L, Miller A, Hartung HP, Overell J, Pei J, Dahlke F, Bernasconi C, Koendgen H, Wang Q, Bonati U, Cohan S. Cognitive effects of ocrelizumab vs interferon beta-1a in relapsing multiple sclerosis: A post hoc analysis of the OPERA I/II trials. Mult Scler Relat Disord. 2025 Mar;95:106310. doi: 10.1016/j.msard.2025.106310. Epub 2025 Feb 2. PMID 39965438
- [Derived] Muros-Le Rouzic E, Heer Y, Yiu S, Tozzi V, Braune S, van Hovell P, Bergmann A, Bernasconi C, Model F, Craveiro L; NTD study group. Five-year efficacy outcomes of ocrelizumab in relapsing multiple sclerosis: A propensity-matched comparison of the OPERA studies with other disease-modifying therapies in real-world lines of treatments. J Cent Nerv Syst Dis. 2024 Sep 13;16:11795735241260563. doi: 10.1177/11795735241260563. eCollection 2024. PMID 39290861
- [Derived] Loomis SJ, Sadhu N, Fisher E, Gafson AR, Huang Y, Yang C, Hughes EE, Marshall E, Herman A, John S, Runz H, Jia X, Bhangale T, Bronson PG. Genome-wide study of longitudinal brain imaging measures of multiple sclerosis progression across six clinical trials. Sci Rep. 2023 Aug 31;13(1):14313. doi: 10.1038/s41598-023-41099-0. PMID 37652990
- [Derived] Kolind S, Gaetano L, Assemlal HE, Bernasconi C, Bonati U, Elliott C, Hagenbuch N, Magon S, Arnold DL, Traboulsee A. Ocrelizumab-treated patients with relapsing multiple sclerosis show volume loss rates similar to healthy aging. Mult Scler. 2023 May;29(6):741-747. doi: 10.1177/13524585231162586. Epub 2023 May 6. PMID 37148240
- [Derived] Laurent SA, Strauli NB, Eggers EL, Wu H, Michel B, Demuth S, Palanichamy A, Wilson MR, Sirota M, Hernandez RD, Cree BAC, Herman AE, von Budingen HC. Effect of Ocrelizumab on B- and T-Cell Receptor Repertoire Diversity in Patients With Relapsing Multiple Sclerosis From the Randomized Phase III OPERA Trial. Neurol Neuroimmunol Neuroinflamm. 2023 Apr 24;10(4):e200118. doi: 10.1212/NXI.0000000000200118. Print 2023 Jul. PMID 37094998
- [Derived] Hauser SL, Bar-Or A, Weber MS, Kletzl H, Gunther A, Manfrini M, Model F, Mercier F, Petry C, Wing Q, Koendgen H, Smith T, Kappos L. Association of Higher Ocrelizumab Exposure With Reduced Disability Progression in Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2023 Feb 15;10(2):e200094. doi: 10.1212/NXI.0000000000200094. Print 2023 Mar. PMID 36792367
- [Derived] Falet JR, Durso-Finley J, Nichyporuk B, Schroeter J, Bovis F, Sormani MP, Precup D, Arbel T, Arnold DL. Estimating individual treatment effect on disability progression in multiple sclerosis using deep learning. Nat Commun. 2022 Sep 26;13(1):5645. doi: 10.1038/s41467-022-33269-x. PMID 36163349
- [Derived] Arnold DL, Sprenger T, Bar-Or A, Wolinsky JS, Kappos L, Kolind S, Bonati U, Magon S, van Beek J, Koendgen H, Bortolami O, Bernasconi C, Gaetano L, Traboulsee A. Ocrelizumab reduces thalamic volume loss in patients with RMS and PPMS. Mult Scler. 2022 Oct;28(12):1927-1936. doi: 10.1177/13524585221097561. Epub 2022 Jun 7. PMID 35672926
- [Derived] Krishnan AP, Song Z, Clayton D, Gaetano L, Jia X, de Crespigny A, Bengtsson T, Carano RAD. Joint MRI T1 Unenhancing and Contrast-enhancing Multiple Sclerosis Lesion Segmentation with Deep Learning in OPERA Trials. Radiology. 2022 Mar;302(3):662-673. doi: 10.1148/radiol.211528. Epub 2021 Dec 14. PMID 34904871
- [Derived] Giovannoni G, Kappos L, de Seze J, Hauser SL, Overell J, Koendgen H, Manfrini M, Wang Q, Wolinsky JS. Risk of requiring a walking aid after 6.5 years of ocrelizumab treatment in patients with relapsing multiple sclerosis: Data from the OPERA I and OPERA II trials. Eur J Neurol. 2022 Apr;29(4):1238-1242. doi: 10.1111/ene.14823. Epub 2021 May 5. PMID 33724637
- [Derived] Hauser SL, Kappos L, Arnold DL, Bar-Or A, Brochet B, Naismith RT, Traboulsee A, Wolinsky JS, Belachew S, Koendgen H, Levesque V, Manfrini M, Model F, Hubeaux S, Mehta L, Montalban X. Five years of ocrelizumab in relapsing multiple sclerosis: OPERA studies open-label extension. Neurology. 2020 Sep 29;95(13):e1854-e1867. doi: 10.1212/WNL.0000000000010376. Epub 2020 Jul 20. PMID 32690791
- [Derived] Kappos L, Wolinsky JS, Giovannoni G, Arnold DL, Wang Q, Bernasconi C, Model F, Koendgen H, Manfrini M, Belachew S, Hauser SL. Contribution of Relapse-Independent Progression vs Relapse-Associated Worsening to Overall Confirmed Disability Accumulation in Typical Relapsing Multiple Sclerosis in a Pooled Analysis of 2 Randomized Clinical Trials. JAMA Neurol. 2020 Sep 1;77(9):1132-1140. doi: 10.1001/jamaneurol.2020.1568. PMID 32511687
- [Derived] Hauser SL, Bar-Or A, Comi G, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Montalban X, Rammohan KW, Selmaj K, Traboulsee A, Wolinsky JS, Arnold DL, Klingelschmitt G, Masterman D, Fontoura P, Belachew S, Chin P, Mairon N, Garren H, Kappos L; OPERA I and OPERA II Clinical Investigators. Ocrelizumab versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):221-234. doi: 10.1056/NEJMoa1601277. Epub 2016 Dec 21. PMID 28002679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1051 participants were screened for entry into study. 821 participants were entered into double-blind treatment period. Participants who completed the 96-week double-blind treatment had option to enter a single group, active treatment open label extension, providing they fulfilled the eligibility criteria and at study completion date, all participants are provided opportunity to rollover and continue treatment and/or safety follow-up under new extension protocol MN43964 (NCT05269004).
Pre-assignment Details: In error, the study completion status for 5 participants in WA21092 was registered as 'Sponsor Termination' in the study eCRF. However, all 5 participants were successfully enrolled into MN43964 and thus have completed the WA21092 study.
Period: Overall Study
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Started | 411 | 410
Entered Open-Label Extension | 326 | 352
Completed | 226 | 239
Not Completed | 185 | 171
Not completed — Death | 6 | 10
Not completed — Physician Decision | 2 | 3
Not completed — Non-compliance with study drug | 3 | 0
Not completed — Lack of Efficacy | 24 | 14
Not completed — Non-compliance | 3 | 2
Not completed — Pregnancy | 5 | 10
Not completed — Protocol Violation | 1 | 1
Not completed — Reason not specified | 42 | 32
Not completed — Consent withdrawn by participant | 41 | 56
Not completed — Adverse Event | 49 | 35
Not completed — Lost to Follow-up | 3 | 6
Not completed — Study Terminated by Sponsor | 4 | 1
Not completed — Missing | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab | Total
Number analyzed (Participants) | 411 | 410 | 821
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (9.3) | 37.1 (9.3) | 37.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 270 | 542
  Male | 139 | 140 | 279

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) in Participants With Relapsing Multiple Sclerosis (MS) at 96 Weeks
Description: ARR was protocol-defined and calculated as the total number of relapses for all participants in the treatment group divided by the total participant-years of exposure to that treatment.
Time Frame: Week 96
Population: Intent-to-treat (ITT) population included all randomized participants in the study.
Measure: Number (95% Confidence Interval); unit: relapses/participant year of treatment
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
relapses/participant year of treatment | 0.292 [0.235 to 0.361] | 0.156 [0.122 to 0.200]
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Adjusted by Geographical Region (US vs. Rest of World) and baseline EDSS (<4.0 vs. >=4.0); Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Rate Ratio = 0.536, 95% CI 2-sided [0.4 to 0.719] — Rate ratio was calculated as Ocrelizumab ARR/Interferon beta-1a 44 mcg SC ARR

2. Secondary Outcome: Time to Onset of Confirmed Disability Progression (CDP) for at Least 12 Weeks During the Double-Blind Treatment Period
Description: Disability progression was defined as an increase in the Expanded Disability Status Scale (EDSS) score of: A) >=1.0 point from the baseline EDSS score when the baseline score was less than or equal to (<=) 5.5 B) >=0.5 point from the baseline EDSS score when the baseline score was >5.5 The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). This outcome measure was considered confirmatory only when results of both studies WA21092 and WA21093 were combined. Disability progression was considered confirmed when the increase in the EDSS was confirmed at a regularly scheduled visit at least 12 weeks after the initial documentation of neurological worsening. EDSS assessment and who were on treatment at time of clinical cut-off date were censored at the date of their last EDSS assessment.
Time Frame: Week 108
Population: ITT population included all randomized participants in the study.
Measure: Median (Full Range); unit: weeks
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
weeks | NA [0 to 103] — Median of time to onset of CDP was not achieved due to low number of participants with events. The full-range values are censored observations. | NA [0 to 108] — Median of time to onset of CDP was not achieved due to low number of participants with events. The full-range values are censored observations.
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Time to onset CDP at week 12; Test type: Superiority or Other; p = 0.0139, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.37 to 0.90]

3. Secondary Outcome: Number of T1 Gadolinium (Gd)-Enhancing Lesions as Detected by Brain Magnetic Resonance Imaging (MRI) During the Double-Blind Treatment
Description: The total number of T1 gadolinium-enhancing lesions for all participants in the treatment group was calculated as the sum of the individual number of lesions at Weeks 24, 48, and 96.
Time Frame: Baseline up to Week 96
Population: ITT population included all randomized participants in the study.
Measure: Number; unit: lesions
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
lesions | 337 | 21
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Adjusted rate ratio = 0.058, 95% CI [0.032 to 0.104] — Adjusted by baseline T1 Gd lesion (present or not), baseline EDSS (<4.0 vs. >=4.0) and geographical region (US vs. rest-of-world). Adjusted rate ratio was calculated as Ocrelizumab adjusted rate/Interferon beta-1a 44 mcg SC adjusted rate

4. Secondary Outcome: Number of New, and/or Enlarging T2 Hyperintense Lesions as Detected by Brain Magnetic Resonance Imaging (MRI) During the Double Blind Treatment
Description: The total number of new and/or enlarging T2 lesions for all participants in the treatment group was calculated as the sum of the individual number of lesions at Weeks 24, 48, and 96.
Time Frame: Baseline up to Week 96
Population: ITT population included all randomized participants in the study.
Measure: Number; unit: lesions
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
lesions | 1916 | 430
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Adjusted rate ratio = 0.229, 95% CI [0.174 to 0.300] — Adjusted by baseline T2 lesion (present or not), baseline EDSS (<4.0 vs. >=4.0) and geographical region (US vs. rest-of-world). Adjusted rate ratio was calculated as Ocrelizumab adjusted rate/Interferon beta-1a 44 mcg SC adjusted rate

5. Secondary Outcome: Percentage of Participants With Confirmed Disability Improvement (CDI) for at Least 12 Weeks
Description: Disability improvement was assessed only for the subgroup of participants with a baseline EDSS score of >= 2.0. It was defined as a reduction in EDSS score of: A) >=1.0 from the baseline EDSS score when the baseline score was >=2 and <=5.5 B) >= 0.5 when the baseline EDSS score > 5.5. The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). This outcome measure was considered confirmatory only when results of both studies WA21092 and WA21093 were combined.
Time Frame: Week 96
Population: ITT population included all randomized participants in the study. Here, number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 306 | 310
percentage of participants | 12.42 [8.94 to 16.64] | 20.00 [15.69 to 24.89]
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.0106, CMH Chi-Squared test (stratified); CMH (Cochran-Mantel-Haenszel) Chi-Squared test Stratified by Geographical Region (US vs. Rest of World) and Baseline EDSS (<4.0 vs. >=4.0); Relative risk (stratified) = 1.61, 95% CI 2-sided [1.11 to 2.33]

6. Secondary Outcome: Time to Onset of Confirmed Disability Progression (CDP) for at Least 24 Weeks During the Double-Blind Treatment Period
Description: Disability progression was defined as an increase in the Expanded Disability Status Scale (EDSS) score of: A) >=1.0 point from the baseline EDSS score when the baseline score was less than or equal to (<=) 5.5 B) >=0.5 point from the baseline EDSS score when the baseline score was >5.5 The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). This outcome measure was considered confirmatory only when results of both studies WA21092 and WA21093 were combined. Disability progression was considered confirmed when the increase in the EDSS was confirmed at a regularly scheduled visit at least 24 weeks after the initial documentation of neurological worsening. Participants who had initial disability progression with no confirmatory EDSS assessment and who were on treatment at time of clinical cut-off date were censored at the date of their last EDSS assessment.
Time Frame: Week 108
Population: ITT population included all randomized participants in the study.
Measure: Median (Full Range); unit: weeks
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
weeks | NA [0 to 103] — Median of time to onset of CDP was not achieved due to low number of participants with events. The full-range values are censored observations. | NA [0 to 108] — Median of time to onset of CDP was not achieved due to low number of participants with events. The full-range values are censored observations.
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Time to onset CDP at week 24; Test type: Superiority or Other; p = 0.0278, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.34 to 0.95]

7. Secondary Outcome: Number of T1 Hypointense Lesions During the Double-Blind Treatment
Description: The total number of new T1-Hypo-Intense Lesions (Chronic Black Holes) for all participants in the treatment group was calculated as the sum of the individual number of new lesions at Weeks 24, 48, and 96.
Time Frame: Baseline up to Week 96
Population: ITT population included all randomized participants in the study.
Measure: Number; unit: lesions
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
lesions | 1307 | 564
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Adjusted rate ratio = 0.428, 95% CI [0.328 to 0.557] — Adjusted by baseline T1-hypointense lesion count, baseline EDSS (<4.0 vs. >=4.0) and geographical region (US vs. rest-of-world). Adjusted rate ratio was calculated as Ocrelizumab adjusted rate/Interferon beta-1a 44 mcg SC adjusted rate

8. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score to Week 96
Description: MSFC score consists of: A) Timed 25-Foot walk; B) 9-Hole Peg Test (9-HPT); and C) Paced Auditory Serial Addition Test (PASAT-3 version). The MSFCS is based on the concept that scores for these three dimensions (arm, leg, and cognitive function) are combined to create a single score (the MSFC) that can be used to detect change over time in a group of participants with MS. Since the three primary measures differ in what they actually measure, a common composite score for the three different measures i.e., Z- score was selected for the purpose. MSFC Score = {Z arm, average + Z leg, average + Z cognitive} / 3.0. The results from each of these three tests are transformed into Z-scores and averaged to yield a composite score for each participant at each time point. A score of +1 indicates that, on average, an individual scored 1 standard deviation (SD) better than the reference population and a score of -1 indicates that an individual scored 1 SD worse than the reference population.
Time Frame: Baseline, Week 96
Population: ITT population included all randomized participants in the study. Here, n signifies the number of participants evaluable at specified time points.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
Z-score
  Unadjusted Baseline mean: number analyzed (Participants) | 359 | 360
  Unadjusted Baseline mean | 0.028 (0.034) | -0.012 (0.040)
  Adjusted Week 96 mean: number analyzed (Participants) | 308 | 322
  Adjusted Week 96 mean | 0.174 (0.031) | 0.213 (0.031)
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.3261, mixed-effect model of repeated measures; Estimates are from analysis based on mixed-effect model of repeated measures (MMRM) using unstructured covariance matrix; Difference in Adjusted Means = 0.039, 95% CI 2-sided [-0.039 to 0.116], Standard Error of Mean 0.039 — Difference in adjusted means was calculated as Ocrelizumab adjusted mean at Week 96/ Interferon beta-1a 44 mcg SC adjusted mean at Week 96

9. Secondary Outcome: Percent Change in Brain Volume as Detected by Brain Magnetic Resonance Imaging (MRI) From Week 24 to Week 96
Description: Brain volume was recorded as an absolute "normalized" value at the baseline visit then recorded at subsequent visits as a percentage change relative to the absolute value at the baseline visit. Therefore, brain volume at Week 24 was calculated as the brain volume at the baseline visit multiplied by 1 + ([percentage change in brain volume from baseline visit to Week 24]/100). Estimates are from analysis based on mixed-effect model of repeated measures (MMRM) using unstructured covariance matrix: Percentage Change = Brain Volume at Week 24 + Geographical Region (US vs. ROW) + Baseline EDSS (< 4.0 vs. >= 4.0) + Week + Treatment + Treatment*Week (repeated values over Week) + Brain Volume at Week 24*Week.
Time Frame: From Week 24 up to Week 96
Population: as for outcome 5
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 267 | 281
percent change | -0.741 (0.046) | -0.572 (0.044)
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.0042, mixed-effect model of repeated measures; [statistical method as in outcome 8, analysis 1]; Difference in Adjusted Means = 0.168, 95% CI 2-sided [0.053 to 0.283], Standard Error of Mean 0.058 — Difference in the rate of brain volume loss: 22.8%. Difference in adjusted means was calculated as Ocrelizumab adjusted mean at Week 96/ Interferon beta-1a 44 mcg SC adjusted mean at Week 96

10. Secondary Outcome: Change From Baseline in Short Form Health Survey-36 (SF-36) Physical Component Summary (PCS) Score at Week 96
Description: The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the PCS and mental composite t-score (MCS). The range for all 8 domains as well as for the composite t- scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Baseline, Week 96
Population: Descriptive statistics at baseline include participants with assessment at baseline and at least one post- baseline value. ITT population included all randomized participants in the study. Here, n signifies the number of participants evaluable at specified time points.
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 411 | 410
t-score
  Unadjusted Baseline mean: number analyzed (Participants) | 338 | 357
  Unadjusted Baseline mean | 45.399 (0.529) | 45.065 (0.507)
  Adjusted mean change at week 96: number analyzed (Participants) | 276 | 315
  Adjusted mean change at week 96 | -0.657 (0.475) | 0.036 (0.456)
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.2193, mixed-effect model of repeated measures; Estimates are from analysis based on mixed-effect model of repeated measures using unstructured covariance matrix; Difference in Adjusted Means = 0.693, 95% CI 2-sided [-0.414 to 1.800], Standard Error of Mean 0.564 — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: Percentage of Participants Who Have No Evidence of Disease Activity (NEDA) up to Week 96
Description: NEDA was defined only for participants with a baseline EDSS score >=2.0. The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Participants who completed the 96- week treatment period were considered as having evidence of disease activity if at least one protocol- defined relapse (PDR), a confirmed disability progression (CDP) event or at least one MRI scan showing MRI activity (defined as Gd-enhancing T1 lesions, or new or enlarging T2 lesions) was reported during the 96-week treatment period, otherwise the participant was considered as having NEDA.
Time Frame: Week 96
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 291 | 289
percentage of participants | 27.1 [22.1 to 32.6] | 47.4 [41.5 to 53.3]
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, CMH Chi-Squared test (stratified); Analyzed using CMH test, stratified by Geographical Region (US vs. rest-of-world) and baseline EDSS (<4.0 vs. >=4.0); Relative risk (stratified) = 1.74, 95% CI 2-sided [1.39 to 2.17]

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs included infusion related reactions (IRRs) and serious MS relapses, but excluded non-serious MS relapses. Serious Adverse Events (SAEs) included serious MS relapses and serious IRRs.
Time Frame: Baseline up to 588 weeks
Population: The safety population included all participants who received any study drug.
Measure: Number; unit: Participants
Groups:
- Interferon Beta-1a + Placebo (Double Blind Period): Interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).
- Ocrelizumab + Placebo (Double Blind Period): Ocrelizumab 600 mg intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week.
- Interferon Beta-1a + Placebo (Open Label Extension); Ocrelizumab + Placebo (Open Label Extension): During the OLE phase, all participants received ocrelizumab 600-mg IV infusion every 24 weeks.
Arm/Group | Interferon Beta-1a + Placebo (Double Blind Period) | Ocrelizumab + Placebo (Double Blind Period) | Interferon Beta-1a + Placebo (Open Label Extension) | Ocrelizumab + Placebo (Open Label Extension)
Number analyzed (Participants) | 409 | 408 | 326 | 352
Participants | 331 | 327 | 302 | 319

13. Secondary Outcome: Exposure to Ocrelizumab (Area Under the Concentration - Time Curve, AUC)
Description: AUC represents total drug exposure for one dosing interval after the 4th dose.
Time Frame: Pre-infusion at Weeks 1, 24, 48, 72; and 30 minutes post-infusion at Week 72; at any time during Weeks 84 and 96
Population: The pharmacokinetics (PK) population included all participants in the ocrelizumab group who had at least 1 measurable concentration value.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter*day
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 393
micrograms per milliliter*day | 3513 (955)

14. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Ocrelizumab
Description: Number of participants positive for anti-drug antibodies (ADAs) to ocrelizumab is the number of post- baseline evaluable participants determined to have treatment-induced ADA or treatment-enhanced ADA during the study period.
Time Frame: Baseline up to week 96
Population: Baseline evaluable participants with an ADA assay result from a baseline sample(s). The safety population included all participants who received any study drug. Here, n signifies the number of participants evaluable at the specified time points.
Measure: Number; unit: Participants
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 409 | 408
Participants
  Positive sample at baseline: number analyzed (Participants) | 397 | 396
  Positive sample at baseline | 2 | 1
  Positive for ADA post-baseline: number analyzed (Participants) | 401 | 402
  Positive for ADA post-baseline | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline to approximately 588 weeks
Description: The safety population includes all enrolled patients who have received at least one dose of any study drug. In the open-label extension (OLE) period, all participants from the double blind period (DBP) had the option to receive ocrelizumab.
Groups:
- Interferon Beta -1a + Placebo (Double Blind Period): Interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).
Arm/Group | Interferon Beta -1a + Placebo (Double Blind Period) | Ocrelizumab + Placebo (Double Blind Period) | Interferon Beta-1a + Placebo (Open Label Extension) | Ocrelizumab + Placebo (Open Label Extension)
All-Cause Mortality (participants affected / at risk) | 1/409 | 0/408 | 6/326 | 11/352
Serious Adverse Events (participants affected / at risk) | 32/409 | 28/408 | 109/326 | 116/352
Other Adverse Events (participants affected / at risk) | 257/409 | 241/408 | 285/326 | 286/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Beta -1a + Placebo (Double Blind Period) (N=409) | Ocrelizumab + Placebo (Double Blind Period) (N=408) | Interferon Beta-1a + Placebo (Open Label Extension) (N=326) | Ocrelizumab + Placebo (Open Label Extension) (N=352)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UVEITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL INCARCERATED HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FUNCTIONAL GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
INTRA-ABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
PEPTIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
GALLBLADDER MUCOCOELE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BILIARY SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 8 (8)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 17 (18) | 20 (23)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DENGUE FEVER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
GENITAL HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES SIMPLEX MENINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTED DERMAL CYST (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTIVE THROMBOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INJECTION SITE CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LYME DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
MASTOIDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
MENINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUROBORRELIOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIORBITAL CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PILONIDAL DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 11 (16) | 6 (7)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST-ACUTE COVID-19 SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SALPINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
SALPINGO-OOPHORITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPTIC ARTHRITIS STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYSTEMIC CANDIDA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUBERCULOSIS BLADDER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUBO-OVARIAN ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE RESPIRATORY FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TENDON DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GLUCOSE TOLERANCE IMPAIRED (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JAW CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL RETROLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THORACIC SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVIX CARCINOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATOFIBROSARCOMA PROTUBERANS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SALIVARY GLAND ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (4) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CERVICAL RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
FACIAL PARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 5 (5)
MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARTIAL SEIZURES WITH SECONDARY GENERALISATION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (3)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANEMBRYONIC GESTATION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CERVICAL INCOMPETENCE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PSYCHOGENIC TREMOR (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABNORMAL UTERINE BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CERVICAL POLYP (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENDOMETRIAL HYPERTROPHY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENITAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MAMMOPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Beta -1a + Placebo (Double Blind Period) (N=409) | Ocrelizumab + Placebo (Double Blind Period) (N=408) | Interferon Beta-1a + Placebo (Open Label Extension) (N=326) | Ocrelizumab + Placebo (Open Label Extension) (N=352)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 22 (25) | 16 (18)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 12 (13) | 19 (22)
FATIGUE (General disorders) | 29 (33) | 21 (22) | 34 (52) | 36 (45)
INFLUENZA LIKE ILLNESS (General disorders) | 85 (97) | 14 (14) | 0 (0) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 73 (75) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 24 (35) | 25 (29)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 46 (65) | 51 (91)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 11 (11) | 19 (26)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 96 (117) | 96 (110)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 21 (25) | 16 (21)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 18 (22) | 16 (25)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 18 (20) | 13 (18)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 30 (33) | 24 (30)
NASOPHARYNGITIS (Infections and infestations) | 40 (52) | 42 (60) | 68 (138) | 73 (156)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 18 (59) | 21 (63)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 17 (20) | 16 (23)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 19 (24) | 15 (15)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 24 (29) | 24 (31)
SINUSITIS (Infections and infestations) | 25 (28) | 18 (22) | 41 (68) | 49 (75)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 35 (44) | 59 (82) | 89 (181) | 90 (182)
URINARY TRACT INFECTION (Infections and infestations) | 56 (81) | 52 (92) | 80 (236) | 101 (296)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 19 (32) | 17 (24)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 31 (47) | 126 (236) | 83 (172) | 71 (179)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 30 (35) | 27 (31) | 46 (57) | 29 (43)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 20 (24) | 24 (27) | 32 (40) | 36 (46)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 19 (24) | 11 (12)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 27 (34) | 24 (34)
HEADACHE (Nervous system disorders) | 54 | 33 | 46 (57) | 40 (47)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 19 (40) | 16 (23)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 (0) | 0 (0) | 82 (163) | 84 (158)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 17 (28) | 18 (23)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 15 (17) | 23 (28)
DEPRESSION (Psychiatric disorders) | 26 (26) | 27 (31) | 24 (28) | 45 (55)
INSOMNIA (Psychiatric disorders) | 15 (15) | 21 (22) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 26 (32) | 30 (46)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 19 (23) | 8 (12)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 23 (24) | 20 (23)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 19 (22) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT01247324/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT01247324/SAP_001.pdf